CLINICAL TRIAL: NCT05267379
Title: An European Multi-centre Cohort Study for Unravelling Pharmacokinetic and Genetic Factors Underlying Post-ERCP Pancreatitis
Acronym: G-PEP
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 108224
Record Dates: First submitted 2022-01-24; First posted 2022-03-04 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PEP patients: Patients who develop PEP
  Interventions: Diagnostic Test: Take blood samples
- Control cohort: Patients who do not develop PEP
  Interventions: Diagnostic Test: Take blood samples

INTERVENTIONS:
Diagnostic Test: Take blood samples — Blood samples are used to check for polymorphisms in NSAID metabolization genes and to determine the diclofenac levels.

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) comes with a risk for post-ERCP pancreatitis (PEP), which accounts for considerable morbidity, high healthcare expenditure, and death. The pathophysiology of PEP and the underpinnings of the preventive effect of rectal NSAID (RN) is poorly understood. Guidelines advise to take preventive measures with a single dose of 100mg RN, peri-ERCP. While NSAID administration reduces the risk with 40%, PEP still occurs after ERCP. In addition, patients with a PEP history have a higher risk to develop recurrence after a subsequent ERCP. This might suggest that an underlying genetic risk may contribute to increasing the incidence of PEP in some patients.

DETAILED DESCRIPTION:
This study is a hypothesis driven and hypothesis free analyses of PEP risk variants. Integrative analysis of NSAID pharmacokinetics and-genetics in PEP patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* written informed consent
* Indication to undergo an ERCP

Exclusion Criteria:

* Pancreatic cancer
* Chronic pancreatitis
* Ongoing acute pancreatitis
* Altered anatomy, defined as anatomical variations in which gall and/or pancreatic juices (in case of pancreatic duct interventions) do not enter the duodenum by way of the ampulla of Vater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with an indication to undergo an ERCP, without pancreatic cancer, chronic pancreatitis, altered anatomy of the upper digestive tract and an ongoing acute pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Differences in SNP's in NSAID metabolization genes | 1 month
  Analyzing differences in polymorphisms in NSAID metabolization genes between PEP patients and control patients using Taqman assay. DNA will be isolated from blood samples and analyzed for SNP's of biotransformation enzymes such as UDP-Glucuronosyltransferase-2B7 (UGT2B7) and CYP2C9. This will be done using polymerase chain reaction (PCR) with fluorescent probes specific for a SNP (Taqman assay)

SECONDARY OUTCOMES:
Diclofenac levels | 2 hours
  Detection of diclofenac levels two hours after diclofenac administration. Levels will be measured in blood samples by high-performance liquid chromatography (HPLC).
Correlation diclofenac levels and NSAID metabolization gene polymorphisms | 1 month
  To investigate whether there is a correlation between diclofenac levels and NSAID metabolism gene polymorphisms. Using an independent t-test, the investigators will try to find a significant correlation between the diclofenac levels and a difference in single nucleotide polymorphism (SNP).
Genes involved in development of PEP | 1 month
  To investigate whether the known genes involved in developing acute pancreatitis also are involved in developing PEP. DNA isolated from the blood samples will be analyzed by Miniseq-technique.

CONTACTS AND LOCATIONS:
Overall Officials: Erwin van Geenen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- RadboudUMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The dataset used during this study is available from the corresponding author upon reasonable request.